CLINICAL TRIAL: NCT02060968
Title: Evaluation of Effectiveness and Safety of Promus PREMIER in Routine Clinical Practice; A Multicenter, Phase-IV, Prospective Observational Study
Brief Title: IRIS-PREMIER REGISTRY
Acronym: IRIS-PREMIER
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Boston Scientific Korea Co. Ltd (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2014-03
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases
Keywords: Promus PREMIER; Routine Clinical Practice
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IRIS PREMIER Cohort: Promus PREMIER
  Interventions: Device: Promus PREMIER

INTERVENTIONS:
Device: Promus PREMIER

SUMMARY:
The purpose of this study is to evaluate effectiveness and safety of Promus PREMIER in Routine Clinical Practice

ELIGIBILITY:
Inclusion Criteria:

* Age 20 and more
* Intervention with Promus PREMIER everolimus eluting coronary stent
* Agreed with written informed consent form

Exclusion Criteria:

* Intervention with Promus PREMIER everolimus eluting coronary stent and other drug eluting stent at the same time
* Life expectancy of 1year and under
* Cardiac shock

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Promus PREMIER stent
Sampling Method: Non-Probability Sample
Enrollment: 2006 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Composite event rate | 1year
  Death, non fatal myocardial infarction, Target Vessel Revascularization

SECONDARY OUTCOMES:
All death | 5year
Cardiac death | 5year
Myocardial infarction | 5year
Composite event of death or myocardial infarction | 5year
Composite event of cardiac death or myocardial infarction | 5year
Target Vessel revascularization | 5year
Target lesion revascularization | 5year
Stent thrombosis by an Academic Research Consortium (ARC) criteria | 5year
Stroke | 5year
Procedural success | 3day
  defined as less than 30% residual stenosis at the completion of procedure without death or Q wave myocardial infarction or urgent revascularization participants will be followed for the duration of hospital stay, an expected average of 3days.

CONTACTS AND LOCATIONS:
Locations (25):
- South Korea (25):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Chungbuk National University Hospital, Cheongju-si
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Gachon University Gil Hospital, Incheon
  - Kwangju Christian Hospital, Kwangju
  - Inje University Pusan Paik Hospital, Pusan
  - Kosin University Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Asan Medical Hospital, Seoul
  - Eulji General Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea St. Paul's Hospital, Seoul
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.